CLINICAL TRIAL: NCT06046547
Title: Integrating Palliative Care Education in Pulmonary Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Centro Hospitalar do Baixo Vouga (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Associate Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PaC/2023
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease
Keywords: Chronic Obstructive Pulmonary Disease; Interstitial Lung Disease; Pulmonary Rehabilitation; Palliative Care; Education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation with palliative care education (Experimental): The experimental group will participate in PR with palliative care education.
  Interventions: Other: Pulmonary rehabilitation integrating education about palliative care
- Pulmonary rehabilitation (Active Comparator): The control group will participate in traditional PR.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation integrating education about palliative care — PR will include exercise training twice a week, and education and psychosocial support once per week during 12 weeks.
  The intervention will include an education session on palliative care, a "Peer-to-peer session", a "Get-apart session" and online sessions.
  The education session on palliative care will be facilitated by two specialist healthcare professionals. The main topics that will be discussed are: concept of palliative care, symptom control, disease impact, psychosocial support and planning for the future.
  Participants will be the primary communicators in the "Peer-to-peer session", and the dialogue will be based on their suggestions. Those who feel more reluctant to reveal private thoughts in front of their loved ones will have the opportunity to discuss their issues in a "Get-apart" environment.
  Individual cases will be referred to a specialist palliative care team or to any other health/social care professional according to the unmet needs identified.
  Arms: Pulmonary rehabilitation with palliative care education
Other: Pulmonary rehabilitation — Participants will receive the same PR program as the experimental group besides the education session on palliative care, the "Peer-to-peer session", the "Get-apart session" and the online sessions (i.e. traditional pulmonary rehabilitation).
  Arms: Pulmonary rehabilitation

SUMMARY:
Living with chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD) imposes enormous daily challenges, especially at advanced stages, not just to patients but also to informal caregivers. Their needs are not fully addressed by disease-modifying treatments. A key strategy to improve their well-being is the early integration of palliative care into routine management of COPD and ILD. Pulmonary rehabilitation (PR), one of the most well-established and cost-effective interventions in chronic respiratory diseases may be a suitable venue for this approach.

The main goal of this randomised controlled study is to explore the effects of palliative care education as part of PR in people with COPD or ILD and informal caregivers. The primary question to be addressed is: "Does integrating education about palliative care in PR improve knowledge on this subject?".

The investigators will compare PR with palliative care education (experimental) with traditional PR (control) in people with COPD or ILD and informal caregivers. The intervention will include an education session about palliative care, a "Peer-to-peer session", a "Get-apart session" and online sessions. A mixed-methods approach will be used to evaluate the outcomes.

This study will provide an evidence-based insight into personalised PR with palliative care education for people with COPD or ILD and informal caregivers.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) and interstitial lung diseases (ILD) have an overwhelming impact on individuals, society and health systems worldwide. Informal caregivers play an essential role in the lives of people with COPD or ILD, however little is known about how to support them. Palliative care addresses multiple unmet needs of people with COPD or ILD and informal caregivers, but it remains highly inaccessible. Pulmonary rehabilitation (PR) is a fundamental evidence-based intervention for the management of COPD and ILD, and may be an opportunity to introduce palliative care. However, the effects of this integrated care model on patients' and informal caregivers' outcomes are still unclear.

Therefore, this study proposes to develop, implement and evaluate an innovative PR model with palliative care education. The primary aim is to explore the effects of palliative care education as part of PR on people with COPD or ILD and informal caregivers' knowledge about palliative care. The secondary aims are: a) to understand the perspectives of people with COPD or ILD and informal caregivers about integrating palliative care education in PR; and b) to explore the short and medium-term effects of palliative care education as part of PR on people with COPD or ILD and informal caregivers' attitude towards palliative care referral, symptoms, disease impact, health-related quality of life (HRQoL), needs, knowledge about the disease and burden.

Recruitment will occur at the outpatient PR unit at Centro Hospitalar Baixo Vouga (CHBV). The pulmonologist of the PR program will identify eligible participants (i.e., people with COPD or ILD and informal caregivers) and explain the study. An appointment for the baseline assessment will be scheduled with those willing to participate.

Participants will be randomised to experimental group (EG) and control group (CG).

Both groups will follow a multidisciplinary team-based PR program, which will include two weekly supervised exercise sessions and weekly education and psychosocial support sessions in a group setting over a 12-week period.

Informal caregivers will be invited to take part in all education and psychosocial support sessions.

The key educational topics explored in the EG group will be: 1) information on chronic respiratory diseases; 2) medication, inhaler techniques, oxygen therapy and non-invasive ventilation; 3) symptom management and exacerbations; 4) palliative care; 5) exercise and physical activity; 6) action plan; 7) anxiety and depression management; and 8) nutrition. Additionally, there will be two sessions: "Peer-to-peer session" and "Get-apart session". In both the focus will be to discuss participants' own issues with the multidisciplinary team. Moreover, every two weeks, participants will have the opportunity to discuss any health-related issue through online sessions.

Individual cases will also be referred for evaluation by a specialist palliative care team or by any other health and social care professional (e.g., psychologist or social worker) according to the specific unmet needs identified.

The EG will receive the PR program as described above and the CG will receive the traditional PR program i.e., without the education session on palliative care, the "Peer-to-peer session", the "Get-apart session" and the online sessions.

Quantitative data will be collected from all participants at baseline, at 12 weeks (i.e., end of PR) and at 6 months post-PR. Qualitative data will be collected only from the EG before and after PR.

The following quantitative data will be collected from people with COPD or ILD: sociodemographic information; health status (e.g., exacerbation(s) within the last 12 months); health literacy; anthropometry; respiratory function; symptoms (pain, dyspnoea, fatigue, cough, and anxiety and depression) and disease impact; HRQoL; needs; functional performance and capacity; peripheral muscle strength; balance; knowledge about palliative care and the disease; and attitude towards palliative care referral.

Informal caregivers will also provide information on: health status (e.g., limitation(s) in activities of daily living); health literacy; role of caring (e.g., relationship with the care receiver); symptoms (pain, fatigue, and anxiety and depression); needs; burden; knowledge about palliative care and the disease; and attitude towards palliative care referral.

Qualitative data will be collected through focus groups. Sample size was estimated with the program G*Power 3.1.9.4, with an effect size specification "as in GPower 3.0", for the within-between interaction of mixed ANOVA with two groups (control and experimental) and two timepoints (pre and post PR). The investigators considered an α of 0.05, a power of 0.80, a correlation among repeated measures of 0.5, a nonsphericity correction of 1 and an expected effect size f of 0.25. The calculated sample size was 34 and considering a possible 40% dropout and missing data rate, the final sample size was determined to be 58.

ELIGIBILITY:
People with COPD or ILD

Inclusion Criteria:

* diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria or multidisciplinary diagnosis of ILD
* clinically stable in the previous month (i.e., without acute exacerbation)

Exclusion Criteria:

* presense of a musculoskeletal, neurological or psychiatric condition which may limit their participation in PR
* participation in any PR program in the last 6 months
* specialist palliative care in the last 12 months
* inability to understand Portuguese

Informal caregivers

Inclusion Criteria:

* adults identified by the participating people with COPD or ILD as informal caregivers; for this purpose, it will be explained to people with COPD or ILD that an informal caregiver is any relative, partner, friend, neighbor, or significant other with personal relationship with them, and who provides a broad range of unpaid assistance, namely with activities of daily living (e.g., toileting, feeding and bathing) and instrumental activities of daily living (e.g., shopping, meal preparation and managing finances)

Exclusion Criteria:

* presense of a neurological or psychiatric condition which may limit their participation
* inability to understand Portuguese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge about palliative care: Palliative Care Knowledge Scale (PaCKS) | Assessment at baseline, at 12-weeks (i.e., end of PR) and at 6 months after PR.
  PaCKS is a 13-item questionnaire assessing a broad range of topics, including goals, target population and timing of palliative care, as well as symptoms and problems that palliative care addresses. For each statement, "True", "False" and "I don't know" options are provided, and a mark is given for each correct answer. Total scores range from 0 to 13 and higher scores indicate higher knowledge.
  It will be evaluated in people with COPD or ILD and informal caregivers.

SECONDARY OUTCOMES:
Attitude towards palliative care referral: "Would you (your loved one) like to be referred to a specialist palliative care team at this time?" | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Possible answers: "Yes", "No" and "I don't know". It will be evaluated in people with COPD or ILD and informal caregivers.
Attitude towards palliative care referral: "Would you (your loved one) like to be referred to a specialist palliative care team if your (your loved one') health deteriorates?" | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Possible answers: "Yes", "No" and "I don't know". It will be evaluated in people with COPD or ILD and informal caregivers who do not answer "Yes" to the previous question.
Pain: "Do you feel pain?" | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Participants will be asked about pain perception with a closed question: "Do you feel pain?". In affirmative cases, pain charts and visual analogue scale will be used to identify its location and to measure its intensity, respectively. Scores will be recorded on a 10 centimetres line that represents a continuum between "no pain" and "worst pain".
  It will be evaluated in people with COPD or ILD and informal caregivers.
Dyspnoea: modified Medical Research Council questionnaire (mMRC) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  mMRC is a 5-point scale graded from 0 ("No breathlessness except on strenuous exercise") to 4 ("Too breathless to leave the house or breathless when dressing or undressing"). Higher scores indicate greater dyspnoea severity on daily activities.
  It will be evaluated in people with COPD or ILD.
Fatigue: Fatigue Functional Assessment of Chronic Illness Therapy-Fatigue Subscale (FACIT-FS) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  FACIT-FS is a 13-item questionnaire assessing tiredness, weakness, listlessness, lack of energy, and their impact on HRQoL. Each item is rated from 0 ("Not at all") to 4 ("Very much"). Total score ranges from 0 to 52. Higher scores indicate less fatigue.
  It will be evaluated in people with COPD or ILD and informal caregivers.
Cough: Leicester Cough Questionnaire (LCQ) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  LCQ is a 19-item questionnaire containing three domains: physical, psychological and social. Each item is rated from 1 to 7. Final score ranges from 3 to 21. Higher scores indicate weaker influence of cough on quality of life.
  It will be evaluated in people with COPD or ILD.
Anxiety and depression: Hospital Anxiety and Depression Scale (HADS) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  HADS includes 14 multiple-choice items divided into 7 item subscales for anxiety (HADS-A) and depression (HADS-D). Scores in each subscale range from 0 to 21. Higher scores indicate greater levels of anxiety and/or depression. Clinically significant anxiety or depression are interpreted by scores ≥8.
  It will be evaluated in people with COPD or ILD and informal caregivers.
Disease impact: COPD Assessment Test (CAT) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  CAT is a 8-item questionnaire which addresses cough, sputum, chest tightness, dyspnoea, home daily activities, confidence leaving home, sleep and energy levels in a 6-point scale rated from 0 to 5. Score ranges from 0 to 40. Higher scores indicate more severe impairment on health status. A score of more than 20 indicates high impact.
  It will be evaluated in people with COPD or ILD.
Health-related quality of life: Saint George's Respiratory Questionnaire (SGRQ) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  SGRQ is a 50-item questionnaire which evaluates three different domains contributing to overall health, daily life, and perceived well-being: symptoms, activity and impact. A score in each domain and a total score are calculated and weighted, ranging from 0 to 100. Higher scores indicate worse HRQoL.
  It will be evaluated in people with COPD or ILD.
Needs: Support Needs Approach for Patients (SNAP) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  SNAP includes 15 questions with the format: "Do you need more support with…" (e.g., "Do you need more support with managing your symptoms?"). For each statement, "No", "A little more" and "Quite a bit more" options are provided to identify the domains in need of support. There is an optional additional open-ended question to capture "anything else" not already covered. The final question refers to the caregiver needs: "Does a family member or friend who helps you need more support?".
  It will be evaluated in people with COPD or ILD.
Needs: Carer Support Needs Assessment Tool (CSNAT) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  CSNAT includes 14 questions covering caregivers' broad support domains which fall into two distinct groups: support that enable them to provide care and more direct personal support for themselves. All questions follow the format: "Do you need more support with…" (e.g., "Do you need more support with knowing what to expect in the future?"). For each question, "No", "A little more", "Quite a bit more" and "Very much more" options are provided to identify support needed within any of the domains. There is an optional additional open-ended question to capture "anything else" not already covered.
  It will be evaluated in informal caregivers.
Functional performance: London Chest Activities of Daily Living (LCADL) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  LCADL includes 15 activities of daily living organized in four domains: self-care, domestic, physical and leisure. Each item is rated from 0 ("I wouldn't do it anyway") to 5 ("I need someone else to do this"), except for one additional question on global impact with "A lot", "A little" and "Not at all" as answer choices. Final score ranges from 0 to 75. Higher scores indicate greater functional limitation.
  It will be evaluated in people with COPD or ILD.
Functional capacity: 6-minute walking test (6-MWT) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  6-MWT evaluates de distance walked at a fast pace during 6 minutes in a 30 meters corridor.
  It will be evaluated in people with COPD or ILD.
Peripheral muscle strength: quadriceps strength, one-repetition maximum (1-RM) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Quadriceps strength, 1-RM: determines the greatest amount of weight that the participant could move in a double leg extension manoeuvre (isotonic strength).
  Measurement is taken on dominant side in kilogram (Kg). It will be evaluated in people with COPD or ILD.
Peripheral muscle strength: handgrip strength, hand-held dynamometer (HHD) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Handgrip strength, HHD: measures the maximum isometric strength of the hand and forearm muscles.
  Measurement is taken on dominant side in kilogram (Kg). It will be evaluated in people with COPD or ILD.
Balance: Brief-Balance Evaluation Systems Test (Brief-BESTest) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Brief-BESTest is 8-item scale evaluating 6 domains contributing to postural control in standing and walking: biomechanical constraints, stability limits/verticality, transitions/anticipatory postural adjustments, reactive postural control, sensory orientation and stability gait. Each domain is evaluated with a test scored from 0 (severe impairment) to 3 (no impairment), with a maximum of 24. Higher scores indicate better balance performance.
  It will be evaluated in people with COPD or ILD.
Knowledge about COPD: Bristol COPD Knowledge Questionnaire (BCKQ) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  BCKQ includes 65 statements divided in 13 topics, each with a stem; these topics cover epidemiology and physiology, aetiology, common symptoms, breathlessness, phlegm, chest infections, exercise, smoking, immunization, inhaled bronchodilators, antibiotics, and oral/inhaled steroids. For each statement, "True", "False" and "I don't know" options are provided, and a mark is given for each correct answer. Total score corresponds to the percentage of correct answers.
  It will be evaluated in people with COPD and informal caregivers.
Burden of providing care: Zarit Burden Interview (ZBI) | Assessment at baseline, at 12-weeks and at 6 months after PR.
  ZBI is a 22-item questionnaire addressing impact of caring experience in several domains: health and wellbeing, personal and social life, and finances. Each question has five response options rated from 0 ("Never") to 4 ("Almost always"), except for the final question on global burden, rated from 0 ("Not at all") to 4 ("Extremely"). Final score ranges from 0 to 88. Higher scores indicate greater burden. A score of more than 24 indicates high burden.
  It will be evaluated in informal caregivers.
Adherence to exercise and education/psychosocial support sessions | Assessment at 12-weeks.
  Adherence to exercise sessions will be evaluated in people with COPD or ILD. Adherence to education and psychosocial support sessions will be evaluated in people with COPD or ILD and informal caregivers.
Occurrence of adverse events | Assessment at 12-weeks.
  Occurrence of adverse events will be evaluated in people with COPD or ILD.
Referral to a specialist palliative care team | Assessment at baseline, at 12-weeks and at 6 months after PR.
  Medical decision to refer a person with COPD or ILD to a specialist palliative care team.

CONTACTS AND LOCATIONS:
Overall Officials: Alda S Marques, PhD, Principal Investigator — Aveiro University
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marx G, Nasse M, Stanze H, Boakye SO, Nauck F, Schneider N. Meaning of living with severe chronic obstructive lung disease: a qualitative study. BMJ Open. 2016 Dec 8;6(12):e011555. doi: 10.1136/bmjopen-2016-011555. PMID 27932338
- [Background] Maddocks M, Lovell N, Booth S, Man WD, Higginson IJ. Palliative care and management of troublesome symptoms for people with chronic obstructive pulmonary disease. Lancet. 2017 Sep 2;390(10098):988-1002. doi: 10.1016/S0140-6736(17)32127-X. PMID 28872031
- [Background] Sigurgeirsdottir J, Halldorsdottir S, Arnardottir RH, Gudmundsson G, Bjornsson EH. COPD patients' experiences, self-reported needs, and needs-driven strategies to cope with self-management. Int J Chron Obstruct Pulmon Dis. 2019 May 16;14:1033-1043. doi: 10.2147/COPD.S201068. eCollection 2019. PMID 31190788
- [Background] Bryant J, Mansfield E, Boyes AW, Waller A, Sanson-Fisher R, Regan T. Involvement of informal caregivers in supporting patients with COPD: a review of intervention studies. Int J Chron Obstruct Pulmon Dis. 2016 Jul 14;11:1587-96. doi: 10.2147/COPD.S107571. eCollection 2016. PMID 27478372
- [Background] Nakken N, Janssen DJ, van den Bogaart EH, Wouters EF, Franssen FM, Vercoulen JH, Spruit MA. Informal caregivers of patients with COPD: Home Sweet Home? Eur Respir Rev. 2015 Sep;24(137):498-504. doi: 10.1183/16000617.00010114. PMID 26324811
- [Background] Miravitlles M, Pena-Longobardo LM, Oliva-Moreno J, Hidalgo-Vega A. Caregivers' burden in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2015 Feb 12;10:347-56. doi: 10.2147/COPD.S76091. eCollection 2015. PMID 25709429
- [Background] Figueiredo D, Gabriel R, Jacome C, Cruz J, Marques A. Caring for relatives with chronic obstructive pulmonary disease: how does the disease severity impact on family carers? Aging Ment Health. 2014;18(3):385-93. doi: 10.1080/13607863.2013.837146. Epub 2013 Sep 20. PMID 24053489
- [Background] Cruz J, Marques A, Figueiredo D. Impacts of COPD on family carers and supportive interventions: a narrative review. Health Soc Care Community. 2017 Jan;25(1):11-25. doi: 10.1111/hsc.12292. Epub 2015 Oct 26. PMID 26499310
- [Background] Giacomini M, DeJean D, Simeonov D, Smith A. Experiences of living and dying with COPD: a systematic review and synthesis of the qualitative empirical literature. Ont Health Technol Assess Ser. 2012;12(13):1-47. Epub 2012 Mar 1. PMID 23074423
- [Background] Figueiredo D, Cruz J, Jacome C, Marques A. Exploring the Benefits to Caregivers of a Family-Oriented Pulmonary Rehabilitation Program. Respir Care. 2016 Aug;61(8):1081-9. doi: 10.4187/respcare.04624. Epub 2016 Jul 5. PMID 27381202
- [Background] Marques A, Jacome C, Cruz J, Gabriel R, Brooks D, Figueiredo D. Family-based psychosocial support and education as part of pulmonary rehabilitation in COPD: a randomized controlled trial. Chest. 2015 Mar;147(3):662-672. doi: 10.1378/chest.14-1488. PMID 25340477
- [Background] Grosbois JM, Gephine S, Kyheng M, Le Rouzic O, Chenivesse C. Improving the wellbeing of caregivers of patients with COPD using a home-based pulmonary rehabilitation programme. ERJ Open Res. 2022 Dec 12;8(4):00255-2022. doi: 10.1183/23120541.00255-2022. eCollection 2022 Oct. PMID 36655219
- [Background] Marques A, Gabriel R, Jacome C, Cruz J, Brooks D, Figueiredo D. Development of a family-based pulmonary rehabilitation programme: an exploratory study. Disabil Rehabil. 2015;37(15):1340-6. doi: 10.3109/09638288.2014.964376. Epub 2014 Sep 25. PMID 25255297
- [Background] Marques A, Cruz J, Brooks D. Interventions to Support Informal Caregivers of People with Chronic Obstructive Pulmonary Disease: A Systematic Literature Review. Respiration. 2021;100(12):1230-1242. doi: 10.1159/000517032. Epub 2021 Jul 14. PMID 34261069
- [Background] Holland AE, Cox NS, Houchen-Wolloff L, Rochester CL, Garvey C, ZuWallack R, Nici L, Limberg T, Lareau SC, Yawn BP, Galwicki M, Troosters T, Steiner M, Casaburi R, Clini E, Goldstein RS, Singh SJ. Defining Modern Pulmonary Rehabilitation. An Official American Thoracic Society Workshop Report. Ann Am Thorac Soc. 2021 May;18(5):e12-e29. doi: 10.1513/AnnalsATS.202102-146ST. PMID 33929307
- [Background] Janssen DJA, Bajwah S, Boon MH, Coleman C, Currow DC, Devillers A, Vandendungen C, Ekstrom M, Flewett R, Greenley S, Guldin MB, Jacome C, Johnson MJ, Kurita GP, Maddocks M, Marques A, Pinnock H, Simon ST, Tonia T, Marsaa K. European Respiratory Society clinical practice guideline: palliative care for people with COPD or interstitial lung disease. Eur Respir J. 2023 Aug 17;62(2):2202014. doi: 10.1183/13993003.02014-2022. Print 2023 Aug. PMID 37290789
- [Background] Reticker AL, Nici L, ZuWallack R. Pulmonary rehabilitation and palliative care in COPD: Two sides of the same coin? Chron Respir Dis. 2012 May;9(2):107-16. doi: 10.1177/1479972312441379. Epub 2012 Apr 12. PMID 22498494
- [Background] Hauser JM, Kramer BJ. Family caregivers in palliative care. Clin Geriatr Med. 2004 Nov;20(4):671-88, vi. doi: 10.1016/j.cger.2004.07.003. PMID 15541619
- [Background] Sullivan DR, Iyer AS, Enguidanos S, Cox CE, Farquhar M, Janssen DJA, Lindell KO, Mularski RA, Smallwood N, Turnbull AE, Wilkinson AM, Courtright KR, Maddocks M, McPherson ML, Thornton JD, Campbell ML, Fasolino TK, Fogelman PM, Gershon L, Gershon T, Hartog C, Luther J, Meier DE, Nelson JE, Rabinowitz E, Rushton CH, Sloan DH, Kross EK, Reinke LF. Palliative Care Early in the Care Continuum among Patients with Serious Respiratory Illness: An Official ATS/AAHPM/HPNA/SWHPN Policy Statement. Am J Respir Crit Care Med. 2022 Sep 15;206(6):e44-e69. doi: 10.1164/rccm.202207-1262ST. PMID 36112774
- [Background] Marques A, Souto-Miranda S, Dias C, Melo E, Jacome C. Access, access, access: the Three A's of pulmonary rehabilitation - perspectives of patients, loved ones and healthcare professionals. ERJ Open Res. 2022 May 3;8(2):00705-2021. doi: 10.1183/23120541.00705-2021. eCollection 2022 Apr. PMID 35509436
- [Background] Seamark DA, Blake SD, Seamark CJ, Halpin DM. Living with severe chronic obstructive pulmonary disease (COPD): perceptions of patients and their carers. An interpretative phenomenological analysis. Palliat Med. 2004 Oct;18(7):619-25. doi: 10.1191/0269216304pm928oa. PMID 15540670
- [Background] Machado A, Almeida S, Burtin C, Marques A. Giving Voice to People - Experiences During Mild to Moderate Acute Exacerbations of COPD. Chronic Obstr Pulm Dis. 2022 Jul 29;9(3):336-348. doi: 10.15326/jcopdf.2022.0283. PMID 35532921
- [Background] Majellano EC, Clark VL, Gibson PG, Foster JM, McDonald VM. The needs and well-being of severe asthma and COPD carers: A cross-sectional study. Respirology. 2022 Feb;27(2):134-143. doi: 10.1111/resp.14167. Epub 2021 Oct 12. PMID 34643011
- [Background] Janssen DJ, McCormick JR. Palliative care and pulmonary rehabilitation. Clin Chest Med. 2014 Jun;35(2):411-21. doi: 10.1016/j.ccm.2014.02.006. Epub 2014 Apr 12. PMID 24874135
- [Derived] Mendes MA, Janssen DJA, Marques A. Integrating palliative care education in pulmonary rehabilitation: a randomized controlled study protocol. BMC Palliat Care. 2024 Mar 20;23(1):76. doi: 10.1186/s12904-024-01363-0. PMID 38504215